CLINICAL TRIAL: NCT02669160
Title: Tolerance of a Motorized Orthosis Reproducing Walking Movement Versus Conventional Passive Standing-up Devices in Children With Cerebral Palsy : A Non-inferiority, Randomised, Multicenter, Controlled Trial
Brief Title: Tolerance of a Motorized Orthosis Reproducing Walking Movement vs Conventional Standing-up Devices in Child With CP
Acronym: EOMEC/CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Collaborators: Région Nord-Pas de Calais, France (Other); Initiatives de parents de Jeunes Epileptiques du Nord (Unknown); Unité de Traitement des Signaux Biomédicaux - HEI (Unknown); Made for Movement (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC-P0032
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: CP (Cerebral Palsy)
Keywords: Motorized Orthotic Devices; Minors; CP (Cerebral Palsy); Exoskeleton Device
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Group of communicating CP children receiving a 30 minutes daily session of verticalization with a motorized orthosis reproducing walking movement (PS Innowalk)
  Interventions: Device: PC Innowalk
- Control (Other): Group of communicating CP children receiving a 30 minutes daily session of verticalization with their conventional passive stander.
  Interventions: Device: Conventional passive stander

INTERVENTIONS:
Device: PC Innowalk
  Arms: Experimental
Device: Conventional passive stander
  Arms: Control

SUMMARY:
Cerebral palsy (CP) includes all the sensorimotor development disorders leading to balance, gait and movement disruptions. These disorders are related to lesions of the central nervous system (CNS) that occurs at birth or during the early childhood. The therapeutic management of CP is essentially based on reeducation, but may also require specific medical treatments, orthopedic devices and sometimes bone surgery. Therefore, CP children are very often placed in specialized institutions with a significant socioeconomic impact. CP children suffer from various sensorimotor impairments, which may evolve into orthopedic deformations, justifying the implementation of restrictive devices. The French High Authority of Health (HAS) estimates that 50 % of CP children have pains when using contention or verticalization devices. These pains are mainly nociceptive and are caused by the passive constraint applied on contact points. Many clinical trials evaluating the physiotherapy benefits on CP patients have led to controversial results regarding the duration of the effect of this therapeutic approach. However, the improvement is more important when neuromuscular facilitation techniques are added to the reeducation program. Human neuronal adaptation and plasticity mechanisms are now understood, with the possibility of a potential partial recovery. Non-invasive stimulation methods and neurorehabilitation techniques could participate in the CNS re-calibration. Automated assisted movements have already been used and these processes showed an increase joint range of motion, bone density and decreased spasticity.

In recent years, "exoskeleton" devices have been used on subjects with spinal cord injuries allowing motor performances improvement.

This pilot study aims evaluating CP children's tolerance to motorized orthosis reproducing walking pattern compared with conventional passive standing-up devices. For this clinical trial, the investigators compare the behavior of CP children using a motorized orthosis reproducing walking pattern (Innowalk Pro Small) to the behavior of same children placed in their usual conventional passive device. The investigators hypothesis is that the Innowalk improves joints range of motion, enhances selective motor control, decreases the medium-term spasticity and offers at least the same tolerance as conventional passive devices.

ELIGIBILITY:
Inclusion Criteria:

* CP children from 6 to 16 years old, and being less than 150 cms, able to receive a 30 minutes verticalization session (standard practice) without sign of discomfort or intolerance
* Communicating children
* Children who had never walked

Exclusion Criteria:

* Children presenting uncontrolled epileptic seizures
* No social insurance affiliation
* Refuse to participate in the study
* Orthopaedic surgery in 6 months which precede the inclusion.
* Injection of botulinum toxin in the 6 months which precede the inclusion.
* Previous neurotomy

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2015-11; Primary Completion 2018-11 (Actual); Study Completion 2018-11-18 (Actual)

PRIMARY OUTCOMES:
Tolerance of pain according to the scale PPP (paediatric pain profile) | 6 weeks
  Paediatric Pain Profile (PPP) pain scale, validated for children with CP and completed by the carer (hetero questionnaire), assessed at D0, D1, W3 and W6.

SECONDARY OUTCOMES:
Lower limb muscular strength measured by the Ashworth scale | 6 weeks
  Ashworth muscle tone scale (assessment of spasticity). This validated scale is used to test the muscular reaction to stretching.
Lower limb articular amplitudes measured by a goniometer | 6 weeks
  Assessment of joint amplitudes using goniometry. This passive assessment will be carried out for the ankle, knee and hip joints.
Selective motor control measured by the CMS/Boyd scale | 6 weeks
  Evaluation of selective motor control using the CMS/Boyd scale.
Stress evaluation measured by the change in heart rate from baseline linked to the verticalization system | 6 weeks
  Heart rate
Identification and quantification (percentage) of adverse events and complications linked to the verticalization system | 6 weeks
  Number of complications (epileptic seizures, lesions, fractures, malaise, etc.) occurring during the study, description of these, severity grade, evolution, responsibility of the equipment, etc
Number of days of utilization of the verticalization system until first complication or withdrawal of the study. | 6 weeks
  Time of use of device until first complication Time in use of device until discontinuation due to complication

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Catanzariti, MD, Principal Investigator — GHICL
Locations (4):
- France (4):
  - IEM Sévigné, Béthune, Hauts-de-France
  - IEM Vent de Bise, Liévin, Hauts-de-France
  - IEM Christian Dabbadie, Villeneuve-d'Ascq, Hauts-de-France
  - IEM Ellen Poidatz, Saint-Fargeau-Ponthierry

IPD SHARING:
Plan to Share IPD: No